CLINICAL TRIAL: NCT00001576
Title: A Phase I Study of Isolated Hepatic Perfusion With Escalating Dose Melphalan Followed by Postoperative Hepatic Arterial Floxuridine and Leucovorin for Metastatic Unresectable Colorectal Cancers of the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970111; 97-C-0111
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-03

CONDITIONS: Colorectal Neoplasm; Liver Neoplasm; Neoplasm Metastasis
Keywords: Regional Therapy; Organ Perfusion; Metastases; Hyperthermia
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis; Hyperthermia | interventions — Melphalan; Floxuridine; Leucovorin

INTERVENTIONS:
Drug: Melphalan
Drug: Floxuridine
Drug: Leucovorin

SUMMARY:
Patients with unresectable metastatic colorectal cancer confined to the liver will undergo a 1 hour hyperthermic isolated hepatic perfusion (IHP) with escalating dose melphalan. Postoperatively, patients will be treated with hepatic arterial infusion of floxuridine (FUDR), 0.2 mg/kg/day and leucovorin (LV), 15 mg/M2/day as a 2-week continuous infusion regimen. Hepatic and systemic toxicity, response to treatment, duration of response, and survival will be followed.

DETAILED DESCRIPTION:
Patients with unresectable metastatic colorectal cancer confined to the liver will undergo a 1 hour hyperthermic isolated hepatic perfusion (IHP) with escalating dose melphalan. Postoperatively, patients will be treated with hepatic arterial infusion of floxuridine (FUDR), 0.2 mg/kg/day and leucovorin (LV), 15 mg/M(2)/day as a 2-week continuous infusion regimen. Hepatic and systemic toxicity, response to treatment, duration of response, and survival will be followed.

ELIGIBILITY:
Histologically or cytologically proven measurable metastatic colorectal cancer limited to the parenchyma of the liver with no evidence of unresectable extrahepatic disease by preoperative radiological studies. Limited resectable extrahepatic disease is acceptable.

Patients must not have been previously treated with intrahepatic artery infusional therapy using FUDR.

Patients mush have had no chemotherapy, radiotherapy or biologic therapy for their malignancy in the month prior to the liver perfusion and must have recovered from all side effects.

Patients must have an ECOG performance standard of 0, 1 or 2 on the day prior to treatment.

Patients must have adequate hepatic function as evidence by bilirubin less than 2.0 and a PT and PTT that are within 1-2 seconds of the upper normal limit.

Patients must not have biopsy proven cirrhosis or evidence of significant portal hypertension by history, endoscopy, or radiologic studies.

Patients must not have a history of congestive heart failure with an LVEF less than 40%.

Patients must not have COPD or other chronic pulmonary disease with PFT's less than 50% predicted for age.

Patients must be 18 years of age or older.

Patients must have a platelet count greater than 100,000 a Hct greater than 27.0, a white blood count greater than 3000/micro liters, and a creatinine less than or equal to 1.5 or a creatinine clearance of greater than 60 ml/min.

Patients must not be pregnant or nursing.

Patients must not be taking immunosuppressive drugs or on chronic anticoagulation.

Patients must not have an active infection.

Patients must not have severe allergic reactions to iodine contrast which can not be controlled by premedication with antihistamines and steroids.

Patients must not have HIV disease.

Patients must be aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks. The patient must be willing to sign an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28
Dates: Start 1997-07; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kemeny N, Conti JA, Cohen A, Campana P, Huang Y, Shi WJ, Botet J, Pulliam S, Bertino JR. Phase II study of hepatic arterial floxuridine, leucovorin, and dexamethasone for unresectable liver metastases from colorectal carcinoma. J Clin Oncol. 1994 Nov;12(11):2288-95. doi: 10.1200/JCO.1994.12.11.2288. PMID 7964942
- [Background] Kemeny N, Seiter K, Conti JA, Cohen A, Bertino JR, Sigurdson ER, Botet J, Chapman D, Mazumdar M, Budd AJ. Hepatic arterial floxuridine and leucovorin for unresectable liver metastases from colorectal carcinoma. New dose schedules and survival update. Cancer. 1994 Feb 15;73(4):1134-42. doi: 10.1002/1097-0142(19940215)73:43.0.co;2-v. PMID 8313315
- [Background] Chang AE, Schneider PD, Sugarbaker PH, Simpson C, Culnane M, Steinberg SM. A prospective randomized trial of regional versus systemic continuous 5-fluorodeoxyuridine chemotherapy in the treatment of colorectal liver metastases. Ann Surg. 1987 Dec;206(6):685-93. doi: 10.1097/00000658-198712000-00001. PMID 2961314